CLINICAL TRIAL: NCT03785522
Title: A Prospective Non-interventional Study Investigating the Treatment Effect of Tresiba® in Adult Patients With Type 2 Diabetes in Saudi Arabia
Brief Title: A Research Study, Looking at How Tresiba® Works in People With Type 2 Diabetes in Local Clinical Practice in Saudi Arabia
Acronym: UPDATES
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4440; U1111-1208-5065 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tresiba®: Patients with type 2 diabetes in Saudi Arabia are to receive Tresiba® (Insulin degludec) for 26 weeks.
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec — Patients will be treated with commercially available Tresiba® in a pre-filled pen injector (FlexTouch®) according to routine clinical practice at the discretion of the study doctor and in accordance with the local label. The study doctor will determine the starting dose of Tresiba® as well as any dose adjustments thereafter.
  Other Names: Tresiba®

SUMMARY:
The purpose of the study is to collect information on how Tresiba® works in real world patients. Patients will get Tresiba® as prescribed to them by their study doctor. The study will last for about 6 to 8 months. Patients will be asked questions about their health and diabetes treatment as part of their normal study doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to initiate treatment with commercially available Tresiba® has been made by the patient/legally acceptable representative and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes and treated with any antihyperglycaemic medication(s), except Tresiba®, for at least 26 weeks prior to Informed consent and Initiation Visit (Visit 1)
* Available and documented HbA1c value measured within the last 12 weeks prior to initiation of Tresiba® treatment

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Hypersensitivity to the active substance or to any of the excipients as specified in the Tresiba® local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes in Saudi Arabia treated with any antihyperglycaemic medication(s), except Tresiba®, are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2018-12-23 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) (percentage) | Week 0 (baseline), Week 26 (end of study)
  Measured in percentage. Baseline is defined as a period of less than or equal to 12 weeks prior to treatment initiation (week 0). If multiple values are available, the most recent one will be used for the baseline. End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in HbA1c (mmol/mol) | Week 0 (baseline), Week 26 (end of study)
  Measured in mmol/mol. Baseline is defined as a period of less than or equal to 12 weeks prior to treatment initiation (week 0). If multiple values are available, the most recent one will be used for the baseline. End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.

SECONDARY OUTCOMES:
Change in fasting plasma glucose (FPG) (mg/dL) | Week 0 (baseline), Week 26 (end of study)
  Measured in mg/dL. Baseline is defined as a period of less than or equal to 12 weeks prior to treatment initiation (week 0). If multiple values are available, the most recent one will be used for the baseline. End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in FPG (mmol/L) | Week 0 (baseline), Week 26 (end of study)
  Measured in mmol/L. Baseline is defined as a period of less than or equal to 12 weeks prior to treatment initiation (week 0). If multiple values are available, the most recent one will be used for the baseline. End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in daily insulin doses: Basal insulin | Week 0 (baseline), Week 26 (end of study)
  Measured in units/day. Baseline dose is defined as the most recent dose prior to treatment initiation (week 0). End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in daily insulin doses: Prandial insulin | Week 0 (baseline), Week 26 (end of study)
  Measured in units/day. Baseline dose is defined as the most recent dose prior to treatment initiation (week 0). End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in daily insulin doses: Total insulin | Week 0 (baseline), Week 26 (end of study)
  Measured in units/day. Baseline dose is defined as the most recent dose prior to treatment initiation (week 0). End of study is defined as the first visit within the window from week 26 to week 34. If multiple values are available for a specific endpoint, the most recent one, relative to the end of study visit will be used.
Change in number of patient reported overall non-severe hypoglycaemic episodes | Week -4 to 0, week 22 to 26
  Number of episodes occurring within 4 weeks prior to initiation of treatment with Tresiba® and within 4 weeks prior to end of study. Non-severe hypoglycaemia is defined as an episode with symptoms and/or self-measured blood glucose (SMBG) value less than or equal to 3.9 mmol/L.
Change in number of patient reported nocturnal non-severe hypoglycaemic episodes | Week -4 to 0, week 22 to 26
  Number of episodes occurring within 4 weeks prior to initiation of treatment with Tresiba® and within 4 weeks prior to end of study. The definition of "nocturnal" will be based on the patient's perception of whether or not it was night, i.e. the answer to this question to the patient: "How many of these occurred between midnight and early morning"?
Change in number of patient reported severe hypoglycaemic episodes (overall) | Week -26 to 0, week 0 to 26
  Number of episodes occurring within 26 weeks prior to initiation of treatment with Tresiba® and within 26 weeks prior to end of study. Severe hypoglycaemia is defined as an episode of hypoglycaemia requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective action. The patient should be asked: "Were you able to treat yourself?", if assistance from another person was required the episode can be defined as severe.
Reason(s) for discontinuing treatment with Tresiba® during the treatment period, if applicable | Week 26
  Pre-specified response option(s) after initiation of treatment with Tresiba® until treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (8):
- Saudi Arabia (8):
  - Novo Nordisk Investigational Site, AL Qateef
  - Novo Nordisk Investigational Site, Dammam
  - Novo Nordisk Investigational Site, Ihsa
  - Novo Nordisk Investigational Site, Jeddah
  - Novo Nordisk Investigational Site, Jubail
  - Novo Nordisk Investigational Site, Khobar
  - Novo Nordisk Investigational Site, Mecca
  - Novo Nordisk Investigational Site, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Derived] AlMalki MH, Aldesokey H, Alkhafaji D, Alsheikh A, Braae UC, Lehrskov LL, Magawry W, Yahia M, Haroun A. Glycaemic Control in People with Type 2 Diabetes Treated with Insulin Degludec: A Real-World, Prospective Non-interventional Study-UPDATES Saudi Arabia. Adv Ther. 2023 Feb;40(2):568-584. doi: 10.1007/s12325-022-02366-0. Epub 2022 Nov 22. PMID 36417058